CLINICAL TRIAL: NCT01803880
Title: A Prospective, Double Blinded, Multicenter, Randomized, Controlled Trial to Evaluate Mechanical Debridement vs. Radiofrequency-Based Debridement in the Treatment of Articular Cartilage Lesions
Brief Title: Mechanical vs. Radiofrequency-Based Debridement in the Treatment of Articular Cartilage Lesions
Acronym: ACT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to meet enrollment goals
Sponsor: Smith & Nephew, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SM-2012-02
Record Dates: First submitted 2013-02-15; First posted 2013-03-04 (Estimated); Results first posted 2019-03-28 (Actual); Last update posted 2019-03-28 (Actual); Status verified 2019-03

CONDITIONS: Chondral Lesion Plus Partial Medial Meniscectomy
Keywords: Articular cartilage; Cartilage lesion; Cartilage defect; Radiofrequency; Debridement; Cartilage; Coblation; Knee; Meniscus; Meniscectomy; MR imaging; Mechanical debridement; Mechanical shaver; Torn meniscus; Arthroscopic knee surgery; Damaged cartilage

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mechanical Debridement (Active Comparator): Mechanical shaver removes areas of damaged tissue
  Interventions: Device: Mechanical Debridement
- RF-based Debridement (Active Comparator): Electrical energy removes areas of damaged tissue (Coblation®)
  Interventions: Device: RF-Based Debridement

INTERVENTIONS:
Device: Mechanical Debridement — mechanical shaver that removes areas of damaged tissue
  Other Names: Mechanical Shaver
  Arms: Mechanical Debridement
Device: RF-Based Debridement — Electrical energy that removes areas of damaged tissue (Coblation®)
  Other Names: Paragon T2 ICW, FLOW 50 wand
  Arms: RF-based Debridement

SUMMARY:
The purpose of this study is to evaluate changes in clinical and imaging outcomes following arthroscopic treatment of a single medial femoral chondral lesion plus partial medial meniscectomy by Radiofrequency-Based debridement or Mechanical Debridement in subjects ≥ eighteen (18) years of age.

DETAILED DESCRIPTION:
This is a non-inferiority, prospective, double blinded, multi-center, randomized, controlled, adaptive study design with enrollment of 82 randomized subjects at up to 13 study sites. Study duration will be until the last subject enrolled reaches 104 weeks post-operative.

The study will be comprised of two parts:

Part I: Part I will require all Investigators perform 1 to 3 procedures using the Quantum 2 Controller plus Paragon T2 ICW Wand or the WEREWOLF Controller plus FLOW 50 Wand. Investigators must be qualified by training to perform procedures prior to use of either study device. This purpose of Part I will be to minimize variability with the recommended directions for use established in the instructions for use (IFU). Part I subjects will be followed per protocol follow-up requirements, and will be included in the safety population only. These subjects will be additive (to the safety population) to the 82 randomized subjects planned as part of the primary evaluation in Part II.

Part II: Part II will consist of 82 randomized subjects. Each Investigator may initiate enrollment of subjects in this part of the study following completion of Part I requirements. The Part II study implements a randomized adaptive study design, whereby an interim analysis will be conducted for sample size re-assessment. There is no intention of reducing the sample size as a result of this interim analysis; however, the sample size may be increased to either establish the non-inferiority and/or may be increased sufficiently to establish superiority depending on the results of the interim analysis.

ELIGIBILITY:
Inclusion Criteria

Subjects MUST meet ALL of the following criteria to be included in the study:

1. Given written informed consent on the IRB/REB approved Consent Form specific to the study, prior to study participation
2. Is male or non pregnant female ≥ eighteen (18) years of age
3. MRI within 9 months of enrollment into this study confirming presence of a medial femoral chondral lesion and medial meniscal tear requiring a partial meniscectomy (as determined by the Investigator)
4. Must present with pain in the index knee of moderate or severe (> 30 mm) as measured by the VAS
5. Must be able to understand English (written and oral)
6. Must be available to come to all study related visits and is physically and mentally willing and able to comply with all post-operative evaluations
7. Must be in general good health (as determined by the Investigator) based on screening assessments and medical history

Intra-operative Inclusion Criteria

Subjects MUST meet ALL of the following criteria to be included in the study:

1. Arthroscopic confirmation of a lesion requiring treatment meeting the following parameters:

1. Single, treatable chondral lesion, localized to the medial femoral condyle,
2. ICRS Grade 2 with widely displaceable fibrillation or flaps or Grade 3A,
3. < 4cm2 in size

Exclusion Criteria

Subjects will be excluded from the study, if they meet ANY one (1) of the following criteria:

1. Body Mass Index (BMI) > 40 or index joint pain is due to BMI (as determined by Investigator)
2. Requires bilateral knee surgery
3. Any of the following conditions:

   1. active joint infections
   2. is immunocompromised, has Sickle Cell disease, has a primary bone disease (e.g., Paget's disease) or disorders that may adversely affect the healing process, or is terminally ill
   3. inflammatory rheumatoid arthritis or other systemic inflammatory arthritis (i.e., gout)
   4. metastatic and/or neoplastic disease
   5. infectious, highly communicable diseases (e.g., active tuberculosis or active hepatitis)
   6. coagulation disorder or patient is receiving anti-coagulants
   7. documented evidence of a history (e.g. liver testing) of drug/alcohol abuse within 12 months of enrollment into this study
   8. diagnosed with a behavioral condition which could affect their ability to accurately comply with the study (e.g. developmental delay, attention deficit disorder, and autism)
4. Any of the following conditions in the index limb or joint:

   1. Grade III or greater osteoarthritis as determined by AP radiograph (Kellgren-Lawrence classification)
   2. systemic steroid therapy or steroid intra-articular therapy within 4 weeks of enrollment into this study
   3. intra-articular viscosupplementation within 3 months of enrollment into this study
   4. osteomyelitis, septicemia, or other infections that may spread to other areas of the body
   5. fractures, osteocysts or osteolysis
   6. recurrent patellar instability (e.g., subluxation or dislocation)
   7. severe Varus or Valgus knee deformities (as determined by Investigator)
   8. symptomatic tear of the lateral meniscus
   9. avascular necrosis
   10. synovial disorders (e.g., pigmented villanodular synovitis)
   11. previous total or partial meniscectomy
   12. requires reconstruction or replacement of medial or lateral meniscus
   13. knee instability, malalignment, or patellar tracking dysfunction
   14. prior treatment for cartilage repair, including but not limited to ACI, Mosaicplasty and/or marrow stimulation procedures
   15. prior knee tendon and/or ligament repair or patellar surgery within 6 months of enrollment into this study
5. Any of the following conditions in the contralateral limb or joint:

   1. greater than minimal abnormality as shown by clinical exam and/or imaging
   2. scheduled or to be scheduled for surgery over the course of this study
   3. involvement causing abnormal ambulation and non-compliance with post-operative rehabilitation guideline
6. The subject has implanted metallic devices (insulin pumps, nerve stimulators, etc), medically implanted clips or other electronically, magnetically or mechanically activated implants that would contraindicate undergoing an MRI scan of the knee
7. The subject has claustrophobia that would inhibit their ability to undergo an MRI scan of the index knee
8. Receiving prescription narcotic pain medication for conditions unrelated to the index knee condition
9. Cardiac pacemaker or other electronic implant(s)
10. Pregnant and/or intending to become pregnant during this study period
11. Participated in a clinical study within 30 days of enrollment into this study, or who is currently participating in another clinical study.
12. Is a prisoner, or is known or suspected to be transient
13. Is involved with Worker's Compensation unrelated to the index knee
14. Is involved with health-related litigation

Intra-operative Exclusion Criteria

Subjects will be excluded from the study, if they meet ANY one (1) of the following criteria:

1. Has more than 1 chondral lesion requiring treatment
2. Requires concomitant procedures (i.e., anterior cruciate ligament repair, high tibial osteotomy), excluding partial medial meniscectomy
3. Has a medial meniscal tear not requiring treatment
4. Has a medial meniscal tear requiring a procedure other than partial meniscectomy
5. Has a lateral meniscal tear requiring treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2013-03-08 (Actual); Primary Completion 2017-05-04 (Actual); Study Completion 2017-07-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jack Farr II, MD, Principal Investigator — Orthopaedic Research Foundation, Inc.; Beate Hansen, MD, PhD, Study Chair — Vice President, Global Clinical Strategy
Locations (7):
- United States (7):
  - Tucson Orthopaedic Institute, Tucson, Arizona
  - Andrews Research and Education Foundation, Inc., Gulf Breeze, Florida
  - Orthopaedic Research Foundation, Inc., Greenwood, Indiana
  - Ohio State University, Columbus, Ohio
  - University Orthopedics Center, State College, Pennsylvania
  - Methodist Center For Orthopedic Surgery, Houston, Texas
  - Basin Orthopedic Surgical Specialists, Odessa, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: There were 148 subjects who initially signed a consent form, although 72 subjects withdrew consent prior to starting the study. This resulted in only 76 subjects actually starting the study and proceeding with study treatment.
Pre-assignment Details: Part I required all qualified investigators to perform 1 to 3 procedures using the study devices for the purpose of minimizing variability with the recommended directions for use established in the instructions for use. Part I subjects were to be included in the safety population only.
Groups:
- Part I: Part I: All Investigators were required to perform 1 to 3 procedures using the study device to minimize variability relating to the technique recommended in the IFU. These subjects were followed per protocol and analyzed for safety findings only.
- Part II: RF-based Debridement: Radiofrequency-Based Debridement was performed using the Quantum 2 Controller plus Paragon T2 ICW Wand or the WEREWOLF Controller plus FLOW 50 Wand. Both systems use a controlled RF-based plasma process (with the trademark 'COBLATION'). In this process, RF energy is used to excite the water molecules in a conductive medium to generate excited radicals within precisely focused plasma. The energized particles in the plasma have sufficient energy to break molecular bonds excising or dissolving (i.e., ablating) soft tissue at relatively low temperatures (typically 40 degrees C to 70 degrees C). The mechanism of action is a chemical process and not a function of the RF energy itself.
- Part II: Mechanical Debridement: Mechanical debridement (i.e., mechanical shaver) was used as the control debridement for the treatment of chondral lesions.
Period: Overall Study
Arm/Group | Part I | Part II: RF-based Debridement | Part II: Mechanical Debridement
Started | 19 | 28 | 29
Completed | 13 | 18 | 14
Not Completed | 6 | 10 | 15
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 4
Not completed — Physician Decision | 0 | 0 | 1
Not completed — Unable to return for follow-up visits | 0 | 1 | 2
Not completed — Lost to Follow-up | 1 | 2 | 3
Not completed — Protocol Violation | 1 | 0 | 0
Not completed — Early study termination | 0 | 6 | 5
Not completed — Incomplete data entry by sites | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part I | Part II: RF-based Debridement | Part II: Mechanical Debridement | Total
Number analyzed (Participants) | 19 | 28 | 29 | 76
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.1 (8.15) | 59.9 (7.22) | 58.0 (9.76) | 57.7 (8.68)
Age, Customized [Count of Participants; unit: Participants]
  Age of Subjects: <40 years | 1 | 0 | 1 | 2
  Age of Subjects: ≥40 years | 18 | 28 | 28 | 74
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 13 | 11 | 32
  Male | 11 | 15 | 18 | 44
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 4 | 6
  Not Hispanic or Latino | 19 | 26 | 25 | 70
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 17 | 27 | 29 | 73
  Black or African American | 2 | 0 | 0 | 2
  Other | 0 | 1 | 0 | 1
  Hispanic | 0 | 1 | 0 | 1
BMI [Mean (Standard Deviation); unit: kg/m^2] | 28.4 (3.02) | 29.9 (3.41) | 29.0 (4.02) | 29.2 (3.57)
Total pre-debridement lesion size [Count of Participants; unit: Participants]
  ≤2 cm^2 | 13 | 19 | 23 | 55
  >2-4 cm^2 | 4 | 9 | 6 | 19
  Missing | 2 | 0 | 0 | 2
Duration (days) since onset of symptoms for index knee [Count of Participants; unit: Participants]
  Acute: ≤30 days | 0 | 3 | 2 | 5
  Subacute: 31 days - 6 months | 8 | 16 | 20 | 44
  Chronic: >6 months | 11 | 9 | 6 | 26
  Missing | 0 | 0 | 1 | 1
Knee Alignment [Count of Participants; unit: Participants]
  Varus malalignment | 1 | 1 | 0 | 2
  Valgus malalignment | 0 | 1 | 0 | 1
  Normal | 18 | 26 | 29 | 73
Narrowest width of meniscal rim post-operatively (radial measurement of meniscus post resection) [Count of Participants; unit: Participants]
  0 - 3º | 5 | 10 | 7 | 22
  >3º | 12 | 18 | 22 | 52
  Missing | 2 | 0 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Knee and Osteoarthritis Outcomes Scores (KOOS) at Week 52 Post-operative
Description: The scores of 5 subscales of KOOS (i.e., Pain, other Symptoms, Function in daily living [ADL], Function in Sport and Recreation [Sport/Rec] and knee related Quality of Life [QoL]) at Baseline, Week 52 and change from Baseline were summarized descriptively by treatment group. The average of KOOS subscale scores was considered as the primary endpoint. For any subject if the value of effectiveness parameter was missing at Week 52 then it was imputed by last observed post-Baseline value (LOCF method).
  Each subscale response is based on a 5-point Likert system with each response score ranging from 0 (no problems) to 4 (extreme problems). Each subscale score is calculated independently. A score of 100 indicated no problems and a score of 0 indicated extreme problems.
  KOOS subscale score = 100 - (mean of the observed items within the subscale x100 / 4)
Time Frame: Postop Week 52
Population: ITT Population
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Part II: RF-based Debridement | Part II: Mechanical Debridement
Number analyzed (Participants) | 28 | 28
score on a scale | 31.94 (3.991) | 39.36 (4.210)
Statistical Analysis 1: Comparison: Part II: RF-based Debridement vs Part II: Mechanical Debridement; An ANCOVA model was used to compare the difference in the devices for change from Baseline in the KOOS at Week 52. KOOS was derived as the average of five subscale scores. LOCF imputation was considered for missing value. One-sided 97.5% confidence interval (CI) for treatment difference (Study-Control) was to be used for determining non-inferiority/superiority of the study device; Test type: Non-Inferiority — Non-inferiority Margin = 10 points. Non-inferiority of study device was concluded if lower limit of one-sided 97.5% CI for treatment difference <10. Superiority of study device was established if LS means of treatment difference and lower limit of one-sided 97.5% CI for treatment difference ≤0; p > 0.05, ANCOVA — All unscheduled visits were to be included and nominal visits were to be applied using analysis visit windows. Both the assigned analysis visits and the site reported nominal visits were provided in the subject data listings; Due to early termination, all inferential analysis was interpreted as descriptive and carried out in an exploratory manner; One-sided 97.5% confidence interval (CI) = -7.42, 97.5% CI 1-sided [lower limit -19.29], Standard Error of Mean 5.137

2. Secondary Outcome: Change in International Knee Documentation Committee (IKDC) Subjective Knee Evaluation Form Scores From Baseline.
Description: The scores of three domains of IKDC Subjective Knee Evaluation Form (i.e., [1] symptoms, including pain, stiffness, swelling, locking/catching, and giving way; [2] sports and daily activities; and [3] current knee function) at Baseline, each of scheduled post-operative visits and changes from Baseline were summarized descriptively by treatment group.
  Change from Baseline in IKDC = IKDC at Baseline + Pseudo-site + Treatment + Treatment*Pseudo-site
  The IKDC score was interpreted by summing the scores for the individual questions and then transforming the score to a scale that ranged from 0 to 100:
  Individual domain IKDC score = [raw score - lowest possible score/range of scores] x 100
  The IKDC total score was interpreted as higher scores = higher function, lower scores = lower function.
  Treatment*Pseudo-site interaction term was non-significant at the 0.05 level and hence was dropped from the statistical method.
Time Frame: Baseline, Postop Weeks 6, 12, 24, 36, 52, and 104/Early Termination (ET)
Population: Not all participants completed the IKDC score questionnaires.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Part II: RF-based Debridement | Part II: Mechanical Debridement
Number analyzed (Participants) | 28 | 29
score on a scale
  IKDC Summary Total Scores (Baseline): number analyzed (Participants) | 28 | 28
  IKDC Summary Total Scores (Baseline) | 39.4 (14.56) | 37.3 (14.40)
  Week 6: number analyzed (Participants) | 27 | 26
  Week 6 | 60.7 (15.42) | 64.4 (16.39)
  Week 6 (Change from Baseline): number analyzed (Participants) | 27 | 26
  Week 6 (Change from Baseline) | 21.0 (13.30) | 27.0 (22.17)
  Week 12: number analyzed (Participants) | 25 | 25
  Week 12 | 69.8 (20.63) | 70.3 (20.24)
  Week 12 (Change from Baseline): number analyzed (Participants) | 25 | 25
  Week 12 (Change from Baseline) | 30.6 (19.57) | 33.1 (20.55)
  Week 24: number analyzed (Participants) | 24 | 22
  Week 24 | 72.9 (21.21) | 70.2 (17.31)
  Week 24 (Change from Baseline): number analyzed (Participants) | 24 | 22
  Week 24 (Change from Baseline) | 33.4 (17.71) | 32.7 (21.07)
  Week 36: number analyzed (Participants) | 20 | 21
  Week 36 | 70.2 (25.61) | 78.8 (15.50)
  Week 36 (Change from Baseline): number analyzed (Participants) | 20 | 21
  Week 36 (Change from Baseline) | 30.6 (22.05) | 41.1 (18.25)
  Week 52: number analyzed (Participants) | 20 | 19
  Week 52 | 75.7 (25.61) | 80.4 (20.26)
  Week 52 (Change from Baseline): number analyzed (Participants) | 20 | 19
  Week 52 (Change from Baseline) | 30.6 (22.05) | 45.3 (21.20)
  Week 104/ET: number analyzed (Participants) | 20 | 14
  Week 104/ET | 77.2 (20.63) | 80.0 (21.66)
  Week 104/ET (Change from Baseline): number analyzed (Participants) | 20 | 14
  Week 104/ET (Change from Baseline) | 36.8 (21.84) | 45.8 (20.46)

3. Secondary Outcome: Number of Participants Stratified by Generalized Laxity Level on IKDC Knee Evaluation
Description: Knee examination with respect to generalized laxity (tight, normal, lax) were summarized as number and percent of subjects in treatment group for Baseline and post-operative follow-up visits.
  The IKDC Knee Evaluation Form was comprised of 3 domains: 1) symptoms including pain, stiffness, swelling, locking/catching, and giving way; 2) sports and daily activities; and 3) current knee function and knee function prior to knee injury.
  There were 18 questions and the raw score was transformed to a 0 to 100 scale score as follows:
  IKDC score = (raw score - lowest possible score / range of scores) x100
Time Frame: Baseline, Postop Weeks 6, 12, 24, 36, 52, and 104/ET
Population: Not all participants completed the IKDC score questionnaires.
Measure: Count of Participants; unit: Participants
Arm/Group | Part II: RF-based Debridement | Part II: Mechanical Debridement
Number analyzed (Participants) | 28 | 29
Participants
  IKDC Score at Baseline - Generalized Laxity: Tight | 0 | 1
  IKDC Score at Baseline - Generalized Laxity: Normal | 28 | 28
  IKDC Score at Baseline - Generalized Laxity: Lax | 0 | 0
  IKDC Score at Week 6 - Generalized Laxity: number analyzed (Participants) | 26 | 26
  IKDC Score at Week 6 - Generalized Laxity: Tight | 0 | 0
  IKDC Score at Week 6 - Generalized Laxity: Normal | 26 | 26
  IKDC Score at Week 6 - Generalized Laxity: Lax | 0 | 0
  IKDC Score at Week 12 - Generalized Laxity: number analyzed (Participants) | 25 | 26
  IKDC Score at Week 12 - Generalized Laxity: Tight | 0 | 0
  IKDC Score at Week 12 - Generalized Laxity: Normal | 25 | 26
  IKDC Score at Week 12 - Generalized Laxity: Lax | 0 | 0
  IKDC Score at Week 24 - Generalized Laxity: number analyzed (Participants) | 24 | 23
  IKDC Score at Week 24 - Generalized Laxity: Tight | 0 | 0
  IKDC Score at Week 24 - Generalized Laxity: Normal | 24 | 23
  IKDC Score at Week 24 - Generalized Laxity: Lax | 0 | 0
  IKDC Score at Week 36 - Generalized Laxity: number analyzed (Participants) | 19 | 22
  IKDC Score at Week 36 - Generalized Laxity: Tight | 0 | 1
  IKDC Score at Week 36 - Generalized Laxity: Normal | 19 | 21
  IKDC Score at Week 36 - Generalized Laxity: Lax | 0 | 0
  IKDC Score at Week 52 - Generalized Laxity: number analyzed (Participants) | 20 | 20
  IKDC Score at Week 52 - Generalized Laxity: Tight | 0 | 0
  IKDC Score at Week 52 - Generalized Laxity: Normal | 20 | 20
  IKDC Score at Week 52 - Generalized Laxity: Lax | 0 | 0
  IKDC Score at Week 104/ET - Generalized Laxity: number analyzed (Participants) | 20 | 15
  IKDC Score at Week 104/ET - Generalized Laxity: Tight | 0 | 0
  IKDC Score at Week 104/ET - Generalized Laxity: Normal | 20 | 15
  IKDC Score at Week 104/ET - Generalized Laxity: Lax | 0 | 0

4. Secondary Outcome: Number of Participants Stratified by Alignment Level on IKDC Knee Evaluation
Description: Knee examination with respect to alignment (obvious varus, normal, obvious valgus) were summarized as number and percent of subjects in treatment group for Baseline and post-operative follow-up visits.
  The IKDC Knee Evaluation Form was comprised of 3 domains: 1) symptoms including pain, stiffness, swelling, locking/catching, and giving way; 2) sports and daily activities; and 3) current knee function and knee function prior to knee injury.
  There were 18 questions and the raw score was transformed to a 0 to 100 scale score as follows:
  IKDC score = (raw score - lowest possible score / range of scores) x100
Time Frame: Baseline, Postop Weeks 6, 12, 24, 36, 52, and 104/ET
Population: Not all participants completed the IKDC score questionnaires.
Measure: Count of Participants; unit: Participants
Arm/Group | Part II: RF-based Debridement | Part II: Mechanical Debridement
Number analyzed (Participants) | 28 | 29
Participants
  IKDC Score at Baseline - Alignment: number analyzed (Participants) | 27 | 29
  IKDC Score at Baseline - Alignment: Obvious Varus | 1 | 0
  IKDC Score at Baseline - Alignment: Normal | 26 | 29
  IKDC Score at Baseline - Alignment: Obvious Valgus | 0 | 0
  IKDC Score at Week 6 - Alignment: number analyzed (Participants) | 26 | 26
  IKDC Score at Week 6 - Alignment: Obvious Varus | 1 | 0
  IKDC Score at Week 6 - Alignment: Normal | 25 | 26
  IKDC Score at Week 6 - Alignment: Obvious Valgus | 0 | 0
  IKDC Score at Week 12 - Alignment: number analyzed (Participants) | 25 | 26
  IKDC Score at Week 12 - Alignment: Obvious Varus | 0 | 1
  IKDC Score at Week 12 - Alignment: Normal | 25 | 25
  IKDC Score at Week 12 - Alignment: Obvious Valgus | 0 | 0
  IKDC Score at Week 24 - Alignment: number analyzed (Participants) | 24 | 23
  IKDC Score at Week 24 - Alignment: Obvious Varus | 0 | 0
  IKDC Score at Week 24 - Alignment: Normal | 24 | 23
  IKDC Score at Week 24 - Alignment: Obvious Valgus | 0 | 0
  IKDC Score at Week 36 - Alignment: number analyzed (Participants) | 19 | 22
  IKDC Score at Week 36 - Alignment: Obvious Varus | 0 | 1
  IKDC Score at Week 36 - Alignment: Normal | 19 | 21
  IKDC Score at Week 36 - Alignment: Obvious Valgus | 0 | 0
  IKDC Score at Week 52 - Alignment: number analyzed (Participants) | 20 | 20
  IKDC Score at Week 52 - Alignment: Obvious Varus | 1 | 0
  IKDC Score at Week 52 - Alignment: Normal | 19 | 20
  IKDC Score at Week 52 - Alignment: Obvious Valgus | 0 | 0
  IKDC Score at Week 104/ET - Alignment: number analyzed (Participants) | 20 | 15
  IKDC Score at Week 104/ET - Alignment: Obvious Varus | 1 | 1
  IKDC Score at Week 104/ET - Alignment: Normal | 19 | 14
  IKDC Score at Week 104/ET - Alignment: Obvious Valgus | 0 | 0

5. Secondary Outcome: Number of Participants Stratified by Patellar Position Level on IKDC Knee Evaluation
Description: Knee examination with respect to patella position (obvious baja, normal, obvious alta) were summarized as number and percent of subjects in treatment group for Baseline and post-operative follow-up visits.
  The IKDC Knee Evaluation Form was comprised of 3 domains: 1) symptoms including pain, stiffness, swelling, locking/catching, and giving way; 2) sports and daily activities; and 3) current knee function and knee function prior to knee injury.
  There were 18 questions and the raw score was transformed to a 0 to 100 scale score as follows:
  IKDC score = (raw score - lowest possible score / range of scores) x100
Time Frame: Baseline, Postop Weeks 6, 12, 24, 36, 52, and 104/ET
Population: Not all participants completed the IKDC score questionnaires.
Measure: Count of Participants; unit: Participants
Arm/Group | Part II: RF-based Debridement | Part II: Mechanical Debridement
Number analyzed (Participants) | 28 | 29
Participants
  IKDC Scores at Baseline - Patella Position: Obvious Baja | 0 | 0
  IKDC Scores at Baseline - Patella Position: Normal | 28 | 29
  IKDC Scores at Baseline - Patella Position: Obvious Alta | 0 | 0
  IKDC Scores at Week 6 - Patella Position: number analyzed (Participants) | 26 | 26
  IKDC Scores at Week 6 - Patella Position: Obvious Baja | 0 | 0
  IKDC Scores at Week 6 - Patella Position: Normal | 26 | 26
  IKDC Scores at Week 6 - Patella Position: Obvious Alta | 0 | 0
  IKDC Scores at Week 12 - Patella Position: number analyzed (Participants) | 25 | 26
  IKDC Scores at Week 12 - Patella Position: Obvious Baja | 0 | 0
  IKDC Scores at Week 12 - Patella Position: Normal | 25 | 26
  IKDC Scores at Week 12 - Patella Position: Obvious Alta | 0 | 0
  IKDC Scores at Week 24 - Patella Position: number analyzed (Participants) | 24 | 23
  IKDC Scores at Week 24 - Patella Position: Obvious Baja | 0 | 0
  IKDC Scores at Week 24 - Patella Position: Normal | 24 | 23
  IKDC Scores at Week 24 - Patella Position: Obvious Alta | 0 | 0
  IKDC Scores at Week 36 - Patella Position: number analyzed (Participants) | 19 | 22
  IKDC Scores at Week 36 - Patella Position: Obvious Baja | 0 | 0
  IKDC Scores at Week 36 - Patella Position: Normal | 19 | 22
  IKDC Scores at Week 36 - Patella Position: Obvious Alta | 0 | 0
  IKDC Scores at Week 52 - Patella Position: number analyzed (Participants) | 20 | 20
  IKDC Scores at Week 52 - Patella Position: Obvious Baja | 0 | 0
  IKDC Scores at Week 52 - Patella Position: Normal | 20 | 20
  IKDC Scores at Week 52 - Patella Position: Obvious Alta | 0 | 0
  IKDC Scores at Week 104/ET - Patella Position: number analyzed (Participants) | 20 | 15
  IKDC Scores at Week 104/ET - Patella Position: Obvious Baja | 0 | 0
  IKDC Scores at Week 104/ET - Patella Position: Normal | 20 | 15
  IKDC Scores at Week 104/ET - Patella Position: Obvious Alta | 0 | 0

6. Secondary Outcome: Number of Participants Stratified by Patella Subluxation/Dislocation Level on IKDC Knee Evaluation
Description: Knee examination with respect to patella subluxation/ dislocation (centered, subluxable, subluxed and dislocated) were summarized as number and percent of subjects in treatment group for Baseline and post-operative follow-up visits.
  The IKDC Knee Evaluation Form was comprised of 3 domains: 1) symptoms including pain, stiffness, swelling, locking/catching, and giving way; 2) sports and daily activities; and 3) current knee function and knee function prior to knee injury.
  There were 18 questions and the raw score was transformed to a 0 to 100 scale score as follows:
  IKDC score = (raw score - lowest possible score / range of scores) x100
Time Frame: Baseline, Postop Weeks 6, 12, 24, 36, 52, and 104/ET
Population: Not all participants completed the IKDC score questionnaires.
Measure: Count of Participants; unit: Participants
Arm/Group | Part II: RF-based Debridement | Part II: Mechanical Debridement
Number analyzed (Participants) | 28 | 29
Participants
  IKDC Scores at Baseline - Subluxation/Dislocation: Centered | 28 | 29
  IKDC Scores at Baseline - Subluxation/Dislocation: Subluxable | 0 | 0
  IKDC Scores at Baseline - Subluxation/Dislocation: Subluxed | 0 | 0
  IKDC Scores at Baseline - Subluxation/Dislocation: Dislocated | 0 | 0
  IKDC Scores at Week 6 - Subluxation/Dislocation: number analyzed (Participants) | 26 | 26
  IKDC Scores at Week 6 - Subluxation/Dislocation: Centered | 26 | 25
  IKDC Scores at Week 6 - Subluxation/Dislocation: Subluxable | 0 | 1
  IKDC Scores at Week 6 - Subluxation/Dislocation: Subluxed | 0 | 0
  IKDC Scores at Week 6 - Subluxation/Dislocation: Dislocated | 0 | 0
  IKDC Scores at Week 12 - Subluxation/Dislocation: number analyzed (Participants) | 25 | 26
  IKDC Scores at Week 12 - Subluxation/Dislocation: Centered | 25 | 26
  IKDC Scores at Week 12 - Subluxation/Dislocation: Subluxable | 0 | 0
  IKDC Scores at Week 12 - Subluxation/Dislocation: Subluxed | 0 | 0
  IKDC Scores at Week 12 - Subluxation/Dislocation: Dislocated | 0 | 0
  IKDC Scores at Week 24 - Subluxation/Dislocation: number analyzed (Participants) | 24 | 23
  IKDC Scores at Week 24 - Subluxation/Dislocation: Centered | 24 | 23
  IKDC Scores at Week 24 - Subluxation/Dislocation: Subluxable | 0 | 0
  IKDC Scores at Week 24 - Subluxation/Dislocation: Subluxed | 0 | 0
  IKDC Scores at Week 24 - Subluxation/Dislocation: Dislocated | 0 | 0
  IKDC Scores at Week 36 - Subluxation/Dislocation: number analyzed (Participants) | 19 | 21
  IKDC Scores at Week 36 - Subluxation/Dislocation: Centered | 19 | 21
  IKDC Scores at Week 36 - Subluxation/Dislocation: Subluxable | 0 | 0
  IKDC Scores at Week 36 - Subluxation/Dislocation: Subluxed | 0 | 0
  IKDC Scores at Week 36 - Subluxation/Dislocation: Dislocated | 0 | 0
  IKDC Scores at Week 52 - Subluxation/Dislocation: number analyzed (Participants) | 20 | 20
  IKDC Scores at Week 52 - Subluxation/Dislocation: Centered | 20 | 20
  IKDC Scores at Week 52 - Subluxation/Dislocation: Subluxable | 0 | 0
  IKDC Scores at Week 52 - Subluxation/Dislocation: Subluxed | 0 | 0
  IKDC Scores at Week 52 - Subluxation/Dislocation: Dislocated | 0 | 0
  IKDC Scores at Week 104/ET - Sublux/Dislocation: number analyzed (Participants) | 20 | 15
  IKDC Scores at Week 104/ET - Sublux/Dislocation: Centered | 20 | 15
  IKDC Scores at Week 104/ET - Sublux/Dislocation: Subluxable | 0 | 0
  IKDC Scores at Week 104/ET - Sublux/Dislocation: Subluxed | 0 | 0
  IKDC Scores at Week 104/ET - Sublux/Dislocation: Dislocated | 0 | 0

7. Secondary Outcome: Change in KOOS Scores From Baseline
Description: The scores of 5 subscales of Knee Injury and Osteoarthritis Outcome Score (KOOS) (i.e., pain, other symptoms, function in daily living [ADL], function in sport and recreation [Sport/Rec], and knee-related Quality of Life [QoL]) change from Baseline were summarized descriptively by treatment group. An ANCOVA model was used to compare the differences in the devices for change from Baseline in the KOOS subscale score at each of the scheduled post-operative visits.
  Each subscale response was based on a 5-point Likert system with each response score ranging from 0 (no problems) to 4 (extreme problems). A score of 100 indicated no problems and a score of 0 indicated extreme problems.
  The KOOS calculations were calculated as follows:
  Individual KOOS subscale scores = 100 - (mean of the observed items within the subscale x100) / 4
  Change from Baseline in KOOS at Week (x) or Day (x) = KOOS at Week (x) or Day (x) - KOOS at Baseline
Time Frame: Baseline, Postop Weeks 6, 12, 24, 36, 52, and 104/ET
Population: Not all participants completed the KOOS questionnaires.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Part II: RF-based Debridement | Part II: Mechanical Debridement
Number analyzed (Participants) | 28 | 29
score on a scale
  Pain - Baseline | 46.2 (17.26) | 50.6 (13.10)
  Pain - Week 6: number analyzed (Participants) | 27 | 27
  Pain - Week 6 | 70.9 (19.62) | 80.4 (14.90)
  Pain - Week 6 (Change from Baseline): number analyzed (Participants) | 27 | 27
  Pain - Week 6 (Change from Baseline) | 25.3 (16.92) | 29.9 (19.66)
  Pain - Week 12: number analyzed (Participants) | 25 | 26
  Pain - Week 12 | 80.6 (20.05) | 82.3 (17.23)
  Pain - Week 12 (Change from Baseline): number analyzed (Participants) | 25 | 26
  Pain - Week 12 (Change from Baseline) | 35.8 (21.92) | 30.3 (19.83)
  Pain - Week 24: number analyzed (Participants) | 24 | 23
  Pain - Week 24 | 78.5 (22.15) | 80.4 (15.39)
  Pain - Week 24 (Change from Baseline): number analyzed (Participants) | 24 | 23
  Pain - Week 24 (Change from Baseline) | 32.5 (21.91) | 29.1 (18.37)
  Pain - Week 36: number analyzed (Participants) | 20 | 22
  Pain - Week 36 | 78.7 (25.98) | 89.0 (9.55)
  Pain - Week 36 (Change from Baseline): number analyzed (Participants) | 20 | 22
  Pain - Week 36 (Change from Baseline) | 29.6 (25.92) | 36.8 (12.94)
  Pain - Week 52: number analyzed (Participants) | 20 | 20
  Pain - Week 52 | 81.5 (24.91) | 87.6 (18.30)
  Pain - Week 52 (Change from Baseline): number analyzed (Participants) | 20 | 20
  Pain - Week 52 (Change from Baseline) | 35.8 (21.98) | 38.2 (18.79)
  Pain - Week 104/ET: number analyzed (Participants) | 20 | 15
  Pain - Week 104/ET | 88.3 (15.18) | 88.5 (17.47)
  Pain - Week 104/ET (Change from Baseline): number analyzed (Participants) | 20 | 15
  Pain - Week 104/ET (Change from Baseline) | 38.9 (21.50) | 39.3 (15.17)
  Other Symptoms - Baseline | 58.4 (20.72) | 54.7 (16.70)
  Other Symptoms - Week 6: number analyzed (Participants) | 27 | 27
  Other Symptoms - Week 6 | 73.5 (17.64) | 75.7 (18.48)
  Other Symptoms - Week 6 (Change from Baseline): number analyzed (Participants) | 27 | 27
  Other Symptoms - Week 6 (Change from Baseline) | 16.0 (20.76) | 20.6 (22.70)
  Other Symptoms - Week 12: number analyzed (Participants) | 25 | 26
  Other Symptoms - Week 12 | 81.3 (19.73) | 83.1 (15.14)
  Other Symptoms - Week 12 (Change from Baseline): number analyzed (Participants) | 25 | 26
  Other Symptoms - Week 12 (Change from Baseline) | 25.0 (25.63) | 28.3 (20.92)
  Other Symptoms - Week 24: number analyzed (Participants) | 24 | 23
  Other Symptoms - Week 24 | 79.8 (20.22) | 80.4 (13.99)
  Other Symptoms - Week 24 (Change from Baseline): number analyzed (Participants) | 24 | 23
  Other Symptoms - Week 24 (Change from Baseline) | 21.9 (22.55) | 25.2 (18.67)
  Other Symptoms - Week 36: number analyzed (Participants) | 20 | 22
  Other Symptoms - Week 36 | 74.1 (23.17) | 87.7 (10.61)
  Other Symptoms - Week 36 (Change from Baseline): number analyzed (Participants) | 20 | 22
  Other Symptoms - Week 36 (Change from Baseline) | 17.0 (24.90) | 31.7 (17.26)
  Other Symptoms - Week 52: number analyzed (Participants) | 20 | 20
  Other Symptoms - Week 52 | 78.7 (24.12) | 88.0 (14.53)
  Other Symptoms - Week 52 (Change from Baseline): number analyzed (Participants) | 20 | 20
  Other Symptoms - Week 52 (Change from Baseline) | 19.8 (26.33) | 34.6 (19.15)
  Other Symptoms - Week 104/ET: number analyzed (Participants) | 20 | 15
  Other Symptoms - Week 104/ET | 83.9 (17.71) | 85.7 (15.57)
  Other Symptoms -Week 104/ET (Change from Baseline): number analyzed (Participants) | 20 | 15
  Other Symptoms -Week 104/ET (Change from Baseline) | 24.5 (23.53) | 34.8 (17.78)
  ADLs - Baseline | 53.5 (21.48) | 57.3 (15.31)
  ADLs - Week 6: number analyzed (Participants) | 27 | 27
  ADLs - Week 6 | 76.6 (21.09) | 86.2 (12.18)
  ADLs - Week 6 (Change from Baseline): number analyzed (Participants) | 27 | 27
  ADLs - Week 6 (Change from Baseline) | 23.3 (18.43) | 29.6 (16.26)
  ADLs - Week 12: number analyzed (Participants) | 25 | 26
  ADLs - Week 12 | 84.1 (21.02) | 85.3 (14.36)
  ADLs - Week 12 (Change from Baseline): number analyzed (Participants) | 25 | 26
  ADLs - Week 12 (Change from Baseline) | 32.0 (24.33) | 27.0 (16.16)
  ADLs - Week 24: number analyzed (Participants) | 24 | 23
  ADLs - Week 24 | 84.6 (20.88) | 87.9 (12.05)
  ADLs - Week 24 (Change from Baseline): number analyzed (Participants) | 24 | 23
  ADLs - Week 24 (Change from Baseline) | 31.1 (24.53) | 31.0 (16.94)
  ADLs - Week 36: number analyzed (Participants) | 20 | 22
  ADLs - Week 36 | 78.7 (23.58) | 91.3 (11.06)
  ADLs - Week 36 (Change from Baseline): number analyzed (Participants) | 20 | 22
  ADLs - Week 36 (Change from Baseline) | 24.3 (24.32) | 32.0 (14.51)
  ADLs - Week 52: number analyzed (Participants) | 20 | 20
  ADLs - Week 52 | 83.6 (23.85) | 89.2 (17.98)
  ADLs - Week 52 (Change from Baseline): number analyzed (Participants) | 20 | 20
  ADLs - Week 52 (Change from Baseline) | 30.4 (24.06) | 32.3 (18.07)
  ADLs - Week 104/ET: number analyzed (Participants) | 20 | 15
  ADLs - Week 104/ET | 89.0 (16.72) | 90.8 (13.39)
  ADLs - Week 104/ET (Change from Baseline): number analyzed (Participants) | 20 | 15
  ADLs - Week 104/ET (Change from Baseline) | 32.6 (24.53) | 36.3 (16.67)
  Sport/Rec - Baseline | 29.9 (22.68) | 30.2 (23.58)
  Sport/Rec - Week 6: number analyzed (Participants) | 27 | 27
  Sport/Rec - Week 6 | 54.1 (25.87) | 61.5 (24.25)
  Sport/Rec - Week 6 (Change from Baseline): number analyzed (Participants) | 27 | 27
  Sport/Rec - Week 6 (Change from Baseline) | 23.1 (27.00) | 29.4 (35.06)
  Sport/Rec - Week 12: number analyzed (Participants) | 25 | 26
  Sport/Rec - Week 12 | 72.0 (24.66) | 67.0 (25.96)
  Sport/Rec - Week 12 (Change from Baseline): number analyzed (Participants) | 25 | 26
  Sport/Rec - Week 12 (Change from Baseline) | 42.3 (30.24) | 38.2 (28.53)
  Sport/Rec - Week 24: number analyzed (Participants) | 24 | 23
  Sport/Rec - Week 24 | 65.6 (30.59) | 69.3 (22.88)
  Sport/Rec - Week 24 (Change from Baseline): number analyzed (Participants) | 24 | 23
  Sport/Rec - Week 24 (Change from Baseline) | 34.9 (32.46) | 40.4 (32.68)
  Sport/Rec - Week 36: number analyzed (Participants) | 20 | 22
  Sport/Rec - Week 36 | 63.0 (33.02) | 75.9 (24.33)
  Sport/Rec - Week 36 (Change from Baseline): number analyzed (Participants) | 20 | 22
  Sport/Rec - Week 36 (Change from Baseline) | 32.8 (35.60) | 45.2 (29.38)
  Sport/Rec - Week 52: number analyzed (Participants) | 20 | 20
  Sport/Rec - Week 52 | 73.0 (30.28) | 78.3 (25.09)
  Sport/Rec - Week 52 (Change from Baseline): number analyzed (Participants) | 20 | 20
  Sport/Rec - Week 52 (Change from Baseline) | 41.4 (30.56) | 51.5 (26.81)
  Sport/Rec - Week 104/ET: number analyzed (Participants) | 20 | 15
  Sport/Rec - Week 104/ET | 76.0 (26.49) | 77.8 (27.88)
  Sport/Rec - Week 104/ET (Change from Baseline): number analyzed (Participants) | 20 | 15
  Sport/Rec - Week 104/ET (Change from Baseline) | 44.2 (25.90) | 53.8 (29.38)
  QoL - Baseline | 28.8 (16.78) | 28.4 (14.90)
  QoL - Week 6: number analyzed (Participants) | 27 | 27
  QoL - Week 6 | 59.7 (21.11) | 59.7 (19.79)
  QoL - Week 6 (Change from Baseline): number analyzed (Participants) | 27 | 27
  QoL - Week 6 (Change from Baseline) | 31.0 (25.09) | 31.3 (26.69)
  QoL - Week 12: number analyzed (Participants) | 25 | 26
  QoL - Week 12 | 66.5 (24.13) | 66.6 (25.55)
  QoL - Week 12 (Change from Baseline): number analyzed (Participants) | 25 | 26
  QoL - Week 12 (Change from Baseline) | 39.0 (27.56) | 37.7 (31.00)
  QoL - Week 24: number analyzed (Participants) | 24 | 23
  QoL - Week 24 | 67.2 (26.98) | 70.7 (21.02)
  QoL - Week 24 (Change from Baseline): number analyzed (Participants) | 24 | 23
  QoL - Week 24 (Change from Baseline) | 36.2 (34.4) | 41.0 (24.70)
  QoL - Week 36: number analyzed (Participants) | 20 | 22
  QoL - Week 36 | 66.3 (32.66) | 77.3 (23.82)
  QoL - Week 36 (Change from Baseline): number analyzed (Participants) | 20 | 22
  QoL - Week 36 (Change from Baseline) | 35.9 (31.86) | 47.4 (25.34)
  QoL - Week 52: number analyzed (Participants) | 20 | 20
  QoL - Week 52 | 72.5 (28.42) | 75.6 (26.59)
  QoL - Week 52 (Change from Baseline): number analyzed (Participants) | 20 | 20
  QoL - Week 52 (Change from Baseline) | 41.9 (25.50) | 47.5 (27.01)
  QoL - Week 104/ET: number analyzed (Participants) | 20 | 15
  QoL - Week 104/ET | 79.1 (21.77) | 76.7 (25.38)
  QoL - Week 104/ET (Change from Baseline): number analyzed (Participants) | 20 | 15
  QoL - Week 104/ET (Change from Baseline) | 46.9 (25.29) | 50.8 (22.89)
  Average KOOS Score - Baseline | 43.4 (17.82) | 44.2 (13.56)
  Average KOOS Score - Week 6: number analyzed (Participants) | 27 | 27
  Average KOOS Score - Week 6 | 67.0 (19.77) | 72.7 (14.47)
  Average KOOS Score - Week 6 (Change from Baseline): number analyzed (Participants) | 27 | 27
  Average KOOS Score - Week 6 (Change from Baseline) | 23.7 (18.85) | 28.2 (20.86)
  Average KOOS Score - Week 12: number analyzed (Participants) | 25 | 26
  Average KOOS Score - Week 12 | 76.9 (20.81) | 76.9 (18.59)
  Average KOOS Score - Week 12 (Change/Baseline): number analyzed (Participants) | 25 | 26
  Average KOOS Score - Week 12 (Change/Baseline) | 34.8 (23.84) | 32.3 (21.05)
  Average KOOS Score - Week 24: number analyzed (Participants) | 24 | 23
  Average KOOS Score - Week 24 | 75.1 (22.69) | 77.8 (15.70)
  Average KOOS Score - Week 24 (Change/Baseline): number analyzed (Participants) | 24 | 23
  Average KOOS Score - Week 24 (Change/Baseline) | 31.3 (23.01) | 33.3 (20.17)
  Average KOOS Score - Week 36: number analyzed (Participants) | 20 | 22
  Average KOOS Score - Week 36 | 71.6 (26.41) | 84.2 (14.59)
  Average KOOS Score - Week 36 (Change/Baseline): number analyzed (Participants) | 20 | 22
  Average KOOS Score - Week 36 (Change/Baseline) | 27.9 (25.78) | 38.6 (16.82)
  Average KOOS Score - Week 52: number analyzed (Participants) | 20 | 20
  Average KOOS Score - Week 52 | 77.9 (25.41) | 83.7 (19.66)
  Average KOOS Score - Week 52 (Change/Baseline): number analyzed (Participants) | 20 | 20
  Average KOOS Score - Week 52 (Change/Baseline) | 33.9 (23.42) | 40.8 (19.97)
  Average KOOS Score - Week 104/ET: number analyzed (Participants) | 20 | 15
  Average KOOS Score - Week 104/ET | 83.3 (17.88) | 83.9 (19.16)
  Average KOOS Score - Week 104/ET (Change/Baseline): number analyzed (Participants) | 20 | 15
  Average KOOS Score - Week 104/ET (Change/Baseline) | 37.4 (21.47) | 43.0 (18.22)

8. Secondary Outcome: Change in Visual Analog Scale (VAS) Scores From Baseline
Description: The VAS knee pain scores were assessed at Baseline, post-operative visits (Day 10, Weeks 6, 12, 24, 36, 52, and 104/ET) and change from Baseline were summarized descriptively by treatment group. An ANCOVA model was used to compare the differences in the devices for change from Baseline in the VAS knee pain score at each of the scheduled post-operative visits. The model had change in VAS knee pain as the response variable and treatment, Baseline VAS knee pain, site, treatment-by-site interaction, lesion-grade, and lesion-grade interaction as independent variables.
  Scores ranged from 0 to 100 with pain intensity measured as none, mild, moderate, or severe:
  No pain (0-4) Mild pain (5-44) Moderate pain (45-74) Severe pain (75-100)
  VAS scores were calculated as:
  Change in VAS knee pain score from Baseline at Week (x) or Day (x) = VAS knee pain at Week (x) or Day (x) - VAS knee pain at Baseline
Time Frame: Baseline, Postop Day 10, Weeks 6, 12, 24, 36, 52, and 104/ET
Population: Not all participants completed the VAS pain score questionnaire.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Part II: RF-based Debridement | Part II: Mechanical Debridement
Number analyzed (Participants) | 28 | 29
units on a scale
  Baseline | 57.6 (19.68) | 59.8 (16.15)
  Day 10 | 28.7 (23.62) | 17.6 (18.69)
  Day 10 (Change from Baseline) | -29.0 (21.29) | -42.2 (23.77)
  Week 6: number analyzed (Participants) | 26 | 26
  Week 6 | 17.8 (23.05) | 13.8 (18.71)
  Week 6 (Change from Baseline): number analyzed (Participants) | 26 | 26
  Week 6 (Change from Baseline) | -38.1 (22.75) | -44.5 (19.90)
  Week 12: number analyzed (Participants) | 25 | 26
  Week 12 | 12.6 (17.71) | 15.2 (17.79)
  Week 12 (Change from Baseline): number analyzed (Participants) | 25 | 26
  Week 12 (Change from Baseline) | -45.8 (23.98) | -41.3 (21.18)
  Week 24: number analyzed (Participants) | 24 | 23
  Week 24 | 15.3 (23.88) | 13.9 (15.38)
  Week 24 (Change from Baseline): number analyzed (Participants) | 24 | 23
  Week 24 (Change from Baseline) | -42.6 (21.98) | -44.2 (18.64)
  Week 36: number analyzed (Participants) | 20 | 22
  Week 36 | 19.1 (26.63) | 7.9 (13.53)
  Week 36 (Change from Baseline): number analyzed (Participants) | 20 | 22
  Week 36 (Change from Baseline) | -37.5 (28.20) | -49.6 (17.18)
  Week 52: number analyzed (Participants) | 20 | 20
  Week 52 | 11.5 (20.08) | 9.3 (19.97)
  Week 52 (Change from Baseline): number analyzed (Participants) | 20 | 20
  Week 52 (Change from Baseline) | -45.8 (20.74) | -49.5 (24.54)
  Week 104/ET: number analyzed (Participants) | 20 | 15
  Week 104/ET | 8.4 (14.22) | 9.9 (20.60)
  Week 104/ET (Change from Baseline): number analyzed (Participants) | 20 | 15
  Week 104/ET (Change from Baseline) | -47.9 (25.92) | -50.7 (30.82)

9. Secondary Outcome: Change in 12-Item Short Form Survey (SF-12) Scores From Baseline - Physical Component Summary (PCS) Score
Description: SF-12 PCS scores at Baseline, post-operative visits (Weeks 6, 12, 24, 36, 52 and 104) and changes from Baseline were summarized descriptively by treatment group. The SF-12 health survey categories included: physical functioning, role functioning physical, bodily pain, general health, vitality, social functioning, role functioning emotional, and mental health. An ANCOVA model was used to compare the difference in the devices for change from Baseline in the SF-12 PCS scores at each of the scheduled post-operative visits. The model had change in SF-12 PCS score as the response variable and treatment, Baseline SF-12 PCS score, site, treatment-by-site interaction, lesion-grade and treatment-by-lesion grade interaction as independent variables.
  Results were expressed as the PCS. Scores could range from 0 (the worst) to 100 (the best).
  SF-12 scores for PCS were calculated as:
  Change in SF-12 PCS score from Baseline at Week (x) = PCS score at Week (x) - PCS score at Baseline
Time Frame: Baseline, Postop Weeks 6, 12, 24, 36, 52, and 104/ET
Population: Not all participants completed the SF-12 questionnaire.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Part II: RF-based Debridement | Part II: Mechanical Debridement
Number analyzed (Participants) | 28 | 29
score on a scale
  Baseline PCS | 36.5 (10.65) | 38.6 (9.63)
  Week 6 PCS: number analyzed (Participants) | 27 | 27
  Week 6 PCS | 45.1 (9.14) | 46.6 (8.27)
  Week 6 PCS (Change from Baseline): number analyzed (Participants) | 27 | 27
  Week 6 PCS (Change from Baseline) | 8.2 (12.62) | 6.7 (9.31)
  Week 12 PCS: number analyzed (Participants) | 25 | 26
  Week 12 PCS | 50.0 (7.87) | 46.6 (8.27)
  Week 12 PCS (Change from Baseline): number analyzed (Participants) | 25 | 26
  Week 12 PCS (Change from Baseline) | 13.4 (13.14) | 9.4 (10.49)
  Week 24 PCS: number analyzed (Participants) | 24 | 23
  Week 24 PCS | 48.5 (9.60) | 50.2 (8.19)
  Week 24 PCS (Change from Baseline): number analyzed (Participants) | 24 | 23
  Week 24 PCS (Change from Baseline) | 11.1 (13.14) | 11.6 (11.12)
  Week 36 PCS: number analyzed (Participants) | 20 | 22
  Week 36 PCS | 46.8 (11.49) | 52.5 (6.98)
  Week 36 PCS (Change from Baseline): number analyzed (Participants) | 20 | 22
  Week 36 PCS (Change from Baseline) | 9.3 (13.81) | 13.1 (10.43)
  Week 52 PCS: number analyzed (Participants) | 19 | 20
  Week 52 PCS | 48.9 (10.24) | 52.5 (8.72)
  Week 52 PCS (Change from Baseline): number analyzed (Participants) | 19 | 20
  Week 52 PCS (Change from Baseline) | 11.6 (10.99) | 14.6 (11.55)
  Week 104/ET PCS: number analyzed (Participants) | 20 | 15
  Week 104/ET PCS | 51.9 (6.96) | 51.6 (8.35)
  Week 104/ET PCS (Change from Baseline): number analyzed (Participants) | 20 | 15
  Week 104/ET PCS (Change from Baseline) | 14.1 (11.02) | 15.3 (11.42)

10. Secondary Outcome: Change in SF-12 Scores From Baseline - Mental Component Summary (MCS) Score
Description: SF-12 MCS scores at Baseline, post-operative visits (Weeks 6, 12, 24, 36, 52, and 104) and changes from Baseline were summarized descriptively by treatment group. The SF-12 health survey categories included: physical functioning, role functioning physical, bodily pain, general health, vitality, social functioning, role functioning emotional, and mental health. An ANCOVA model was used to compare the difference in the devices for change from Baseline in the SF-12 MCS scores at each of the scheduled post-operative visits. The model had change in SF-12 MCS score as the response variable and treatment, Baseline SF-12 MCS score, site, treatment-by-site interaction, lesion-grade and treatment-by-lesion grade interaction as independent variables.
  Results were expressed as the MCS. Scores could range from 0 (the worst) to 100 (the best).
  SF-12 scores for MCS were calculated as:
  Change in SF-12 MCS score from Baseline at Week (x) = MCS score at Week (x) - MCS score at Baseline
Time Frame: Baseline, Postop Weeks 6, 12, 24, 36, 52, and 104/ET
Population: Not all participants completed the SF-12 questionnaire.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Part II: RF-based Debridement | Part II: Mechanical Debridement
Number analyzed (Participants) | 28 | 29
score on a scale
  Baseline MCS | 55.9 (9.98) | 55.1 (9.52)
  Week 6 MCS: number analyzed (Participants) | 27 | 27
  Week 6 MCS | 55.1 (8.44) | 57.5 (9.63)
  Week 6 MCS (Change from Baseline): number analyzed (Participants) | 27 | 27
  Week 6 MCS (Change from Baseline) | -0.1 (8.87) | 3.4 (8.27)
  Week 12 MCS: number analyzed (Participants) | 25 | 26
  Week 12 MCS | 55.6 (7.47) | 55.9 (7.75)
  Week 12 MCS (Change from Baseline): number analyzed (Participants) | 25 | 26
  Week 12 MCS (Change from Baseline) | 0.5 (10.97) | 1.2 (8.05)
  Week 24 MCS: number analyzed (Participants) | 24 | 23
  Week 24 MCS | 56.6 (5.32) | 56.9 (8.47)
  Week 24 MCS (Change from Baseline): number analyzed (Participants) | 24 | 23
  Week 24 MCS (Change from Baseline) | 0.7 (10.17) | 2.6 (8.32)
  Week 36 MCS: number analyzed (Participants) | 20 | 22
  Week 36 MCS | 55.5 (6.49) | 57.1 (4.81)
  Week 36 MCS (Change from Baseline): number analyzed (Participants) | 20 | 22
  Week 36 MCS (Change from Baseline) | 0.1 (10.63) | 1.8 (7.61)
  Week 52 MCS: number analyzed (Participants) | 19 | 20
  Week 52 MCS | 56.1 (7.19) | 56.1 (4.90)
  Week 52 MCS (Change from Baseline): number analyzed (Participants) | 19 | 20
  Week 52 MCS (Change from Baseline) | 0.6 (9.46) | 1.5 (10.35)
  Week 104/ET MCS: number analyzed (Participants) | 20 | 15
  Week 104/ET MCS | 56.1 (5.17) | 55.7 (9.91)
  Week 104/ET MCS (Change from Baseline): number analyzed (Participants) | 20 | 15
  Week 104/ET MCS (Change from Baseline) | -0.4 (10.84) | 0.1 (10.54)

11. Secondary Outcome: Change in EuroQoL 5 Dimensions, 5 Level Scale (EQ-5D-5L) Scores From Baseline (EQ-5D-5L Summary Total Score)
Description: The EQ-5D-5L and EQ-VAS surveys were assessed at the specified time points. The EQ-5D-5L score was composed of 5 dimensions to assess mobility, self-care, usual activities, pain/discomfort, and anxiety/depression based on participant's responses. Each individual category calculated a score of between -1 and +1. A score of -1 showed the worst improvement and a score of +1 showed the most improvement.
  Summary total scores for EQ-5D-5L were calculated as:
  Change in EQ-5D-5L score from Baseline at Week (x) or Day (x) = EQ-5D-5L score at Week (x) or Day (x) - EQ-5D-5L score at Baseline
Time Frame: Baseline, Postop Day 10, Weeks 6, 12, 24, 36, 52, and 104/ET
Population: Not all participants completed the EQ-5D-5L questionnaire.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Part II: RF-based Debridement | Part II: Mechanical Debridement
Number analyzed (Participants) | 28 | 29
units on a scale
  EQ-5D-5L Summary Total Score (Baseline) | 0.714 (0.1503) | 0.745 (0.910)
  Day 10 | 0.738 (0.1309) | 0.788 (0.0967)
  Day 10 (Change from Baseline) | 0.024 (0.1331) | 0.043 (0.1151)
  Week 6: number analyzed (Participants) | 26 | 26
  Week 6 | 0.791 (0.1528) | 0.825 (0.0999)
  Week 6 (Change from Baseline): number analyzed (Participants) | 26 | 26
  Week 6 (Change from Baseline) | 0.083 (0.1080) | 0.081 (0.1318)
  Week 12: number analyzed (Participants) | 25 | 26
  Week 12 | 0.823 (0.1614) | 0.854 (0.1145)
  Week 12 (Change from Baseline): number analyzed (Participants) | 25 | 26
  Week 12 (Change from Baseline) | 0.116 (0.1182) | 0.094 (0.1137)
  Week 24: number analyzed (Participants) | 24 | 23
  Week 24 | 0.814 (0.1473) | 0.854 (0.1047)
  Week 24 (Change from Baseline): number analyzed (Participants) | 24 | 23
  Week 24 (Change from Baseline) | 0.100 (0.1436) | 0.105 (0.1269)
  Week 36: number analyzed (Participants) | 20 | 22
  Week 36 | 0.806 (0.1650) | 0.914 (0.0895)
  Week 36 (Change from Baseline): number analyzed (Participants) | 20 | 22
  Week 36 (Change from Baseline) | 0.096 (0.1524) | 0.143 (0.0743)
  Week 52: number analyzed (Participants) | 20 | 20
  Week 52 | 0.835 (0.1950) | 0.911 (0.1267)
  Week 52 (Change from Baseline): number analyzed (Participants) | 20 | 20
  Week 52 (Change from Baseline) | 0.135 (0.1502) | 0.162 (0.1362)
  Week 104/ET: number analyzed (Participants) | 20 | 15
  Week 104/ET | 0.843 (0.1290) | 0.906 (0.1298)
  Week 104/ET (Change from Baseline): number analyzed (Participants) | 20 | 15
  Week 104/ET (Change from Baseline) | 0.106 (0.1381) | 0.167 (0.1470)

12. Secondary Outcome: Change in EQ-5D-5L Scores From Baseline (EQ-VAS Summary Total Score)
Description: The EQ-5D-5L and EQ-VAS surveys were assessed at the specified time points. The EQ-5D-5L score was composed of 5 dimensions to assess mobility, self-care, usual activities, pain/discomfort, and anxiety/depression based on participant's responses.
  The EQ-VAS score ranged from 0 to 100 with higher scores representing better health and lower scores representing worse health.
  Summary total scores for EQ-VAS were calculated as:
  Change in EQ-VAS score from Baseline at Week (x) or Day (x) = EQ-VAS score at Week (x) or Day (x) - EQ-VAS score at Baseline
Time Frame: Baseline, Postop Day 10, Weeks 6, 12, 24, 36, 52, and 104/ET
Population: Not all participants completed the EQ-VAS questionnaire.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Part II: RF-based Debridement | Part II: Mechanical Debridement
Number analyzed (Participants) | 28 | 29
score on a scale
  EQ-VAS Summary Total Score (Baseline) | 74.9 (21.70) | 76.3 (17.90)
  Day 10 | 80.7 (16.85) | 88.0 (8.87)
  Day 10 (Change from Baseline) | 5.8 (18.42) | 11.7 (16.80)
  Week 6: number analyzed (Participants) | 26 | 26
  Week 6 | 84.0 (13.99) | 89.5 (7.41)
  Week 6 (Change from Baseline): number analyzed (Participants) | 26 | 26
  Week 6 (Change from Baseline) | 10.5 (14.82) | 14.1 (17.87)
  Week 12: number analyzed (Participants) | 25 | 26
  Week 12 | 84.6 (14.35) | 90.1 (7.06)
  Week 12 (Change from Baseline): number analyzed (Participants) | 25 | 26
  Week 12 (Change from Baseline) | 10.8 (13.11) | 14.3 (18.55)
  Week 24: number analyzed (Participants) | 24 | 23
  Week 24 | 87.3 (12.97) | 88.4 (10.98)
  Week 24 (Change from Baseline): number analyzed (Participants) | 24 | 23
  Week 24 (Change from Baseline) | 13.3 (16.09) | 14.0 (16.63)
  Week 36: number analyzed (Participants) | 20 | 22
  Week 36 | 84.7 (12.97) | 91.0 (6.01)
  Week 36 (Change from Baseline): number analyzed (Participants) | 20 | 22
  Week 36 (Change from Baseline) | 13.3 (16.09) | 15.0 (17.81)
  Week 52: number analyzed (Participants) | 20 | 20
  Week 52 | 84.1 (18.50) | 90.2 (8.60)
  Week 52 (Change from Baseline): number analyzed (Participants) | 20 | 20
  Week 52 (Change from Baseline) | 8.6 (18.55) | 15.1 (17.24)
  Week 104/ET: number analyzed (Participants) | 20 | 15
  Week 104/ET | 87.1 (12.96) | 90.3 (11.55)
  Week 104/ET (Change from Baseline): number analyzed (Participants) | 20 | 15
  Week 104/ET (Change from Baseline) | 9.2 (13.04) | 14.9 (13.27)

13. Secondary Outcome: Subject Satisfaction Postoperatively at Weeks 52 and 104
Description: Subjects were questioned regarding their satisfaction with study treatment for knee pain.
Time Frame: Postop Weeks 52 and 104/ET
Population: Not all participants completed the subject satisfaction questionnaire.
Measure: Count of Participants; unit: Participants
Arm/Group | Part II: RF-based Debridement | Part II: Mechanical Debridement
Number analyzed (Participants) | 29 | 29
Participants
  Week 52: number analyzed (Participants) | 19 | 20
  Week 52: Extremely Satisfied | 0 | 0
  Week 52: Very Satisfied | 12 | 16
  Week 52: Somewhat Satisfied | 5 | 2
  Week 52: Somewhat Dissatisfied | 2 | 2
  Week 52: Very Dissatisfied | 0 | 0
  Week 52: Extremely Dissatisfied | 0 | 0
  Week 104/ET: number analyzed (Participants) | 20 | 15
  Week 104/ET: Extremely Satisfied | 0 | 0
  Week 104/ET: Very Satisfied | 15 | 13
  Week 104/ET: Somewhat Satisfied | 5 | 2
  Week 104/ET: Somewhat Dissatisfied | 0 | 0
  Week 104/ET: Very Dissatisfied | 0 | 0
  Week 104/ET: Extremely Dissatisfied | 0 | 0

14. Secondary Outcome: Magnetic Resonance Imaging (MRI) and International Cartilage Repair Society (ICRS) Chondral Lesion Assessments
Description: MRIs were obtained post-operatively at Day 10, obtained during the time period of Day 10 through Week 52, and again obtained during the time period of Week 52 through Week 104/ET). The images were evaluated using ICRS assessments of chondral lesions to determine the percentage of change in cartilage lesions over time post-operatively.
  ICRS partial-thickness chondral lesion assessment scores:
  Low-grade defect = less than 50% High-grade defect = 50% to 99%
Time Frame: Postop Day 10, Day 10 to Week 52, Week 52 to Week 104/ET
Population: Only Baseline subjects and subjects showing a percentage change in cartilage signal were included in the imaging results.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Part I | Part II: RF-based Debridement | Part II: Mechanical Debridement
Number analyzed (Participants) | 19 | 28 | 29
units on a scale
  Postop Day 10 (Baseline) - Percent (%) Lesion Fill: number analyzed (Participants) | 17 | 28 | 27
  Postop Day 10 (Baseline) - Percent (%) Lesion Fill | 50.5 (15.5) | 52.9 (16.6) | 53.5 (16.8)
  Day 10 to Week 52 - <50% Change in Lesion Fill: number analyzed (Participants) | 6 | 6 | 7
  Day 10 to Week 52 - <50% Change in Lesion Fill | -0.3 (8.1) | -1.9 (4.4) | 1.5 (6.6)
  Day 10 to Week 52 - ≥50% Change in Lesion Fill: number analyzed (Participants) | 8 | 12 | 11
  Day 10 to Week 52 - ≥50% Change in Lesion Fill | 1.2 (11.1) | -3.4 (5.9) | -5.5 (10.8)
  Weeks 52 to 104/ET - <50% Change in Lesion Fill: number analyzed (Participants) | 5 | 3 | 4
  Weeks 52 to 104/ET - <50% Change in Lesion Fill | -5.2 (13.4) | 2.9 (8.8) | -6.0 (11.9)
  Weeks 52 to 104/ET - ≥50% Change in Lesion Fill: number analyzed (Participants) | 7 | 9 | 7
  Weeks 52 to 104/ET - ≥50% Change in Lesion Fill | 1.2 (14.7) | -3.4 (8.6) | 3.7 (4.7)

ADVERSE EVENTS:
Time Frame: AEs were recorded from the time of surgery until subject completion, ET, or study termination, whichever happened first, assessed throughout the 24-month follow-up period.
Arm/Group | Part I | Part II: RF-based Debridement | Part II: Mechanical Debridement
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/28 | 0/29
Serious Adverse Events (participants affected / at risk) | 1/19 | 2/28 | 1/29
Other Adverse Events (participants affected / at risk) | 13/19 | 26/28 | 19/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part I (N=19) | Part II: RF-based Debridement (N=28) | Part II: Mechanical Debridement (N=29)
Hernia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Patella fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part I (N=19) | Part II: RF-based Debridement (N=28) | Part II: Mechanical Debridement (N=29)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (10) | 20 (27) | 13 (14) — Note: only 1 reported event of Arthralgia was assessed as related to study device.
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
VIIth nerve paralysis (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 2 (2)
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 1 (1) | 0 (0)
Hernia Pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) | 2 (2)
Blood pressure increased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 2 (2)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Joint effusion (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 1 (1)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Due to early termination of the study, all inferential analyses were noted as descriptive and the clinical outcome results should be interpreted with caution.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Authorship and contents of publications shall be discussed between each Principal Investigator and Sponsor. Sponsor shall serve as coordinator of multi-center study disclosures and, in event of a disagreement among investigators, Sponsor shall determine resolution of any such dispute. Sponsor shall be furnished copies of any proposed multi-center publication or disclosure at least 90 days prior to the proposed date for submission for publication or disclosure.

DOCUMENTS (2):
  • Study Protocol (2016-10-27): https://cdn.clinicaltrials.gov/large-docs/80/NCT01803880/Prot_000.pdf
  • Statistical Analysis Plan (2017-03-10): https://cdn.clinicaltrials.gov/large-docs/80/NCT01803880/SAP_001.pdf